CLINICAL TRIAL: NCT04773275
Title: INCITE LS: A Clinical Evaluation of the Aliya™ System in Late Stage Cancer
Brief Title: A Clinical Evaluation of the Aliya™ System in Late Stage Cancer
Acronym: INCITE LS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Galvanize Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-00010
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cancer of Lung, Kidney or Liver
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Single cohort consecutive case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Aliya PEF treatment (Experimental)
  Interventions: Device: Pulsed electric field treatment using the Aliya system

INTERVENTIONS:
Device: Pulsed electric field treatment using the Aliya system — Patients will undergo pulsed electric field (PEF) treatment of up to 5 tumors (new or progressing) measuring ≤ 2cm in longest diameter.

SUMMARY:
A prospective, single-arm, non-randomized, multi-center, open-label study following patients to 1 year. The study is designed to evaluate the safety and clinical utility of Pulsed Electric Field (PEF) treatment of advanced stage or metastatic cancer following progression on immunotherapy.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and clinical utility of Pulsed Electric Field (PEF) treatment of advanced stage or metastatic cancer following progression on immunotherapy. The study will enroll adult patients with confirmed 8th ed. Stage IV non-small cell lung cancer (NSCLC), Stage IV renal cell carcinoma (RCC), or Stage IV hepatocellular carcinoma (HCC), who have experienced a response to checkpoint inhibitor (CPI) therapy (complete response (CR), partial response (PR), or stable disease (SD) as per RECIST 1.1) for a minimum of 6 months, and have documented radiologic progression (progressive disease (PD) as defined by RECIST 1.1) in up to five sites (non-central nervous system). PEF treatment delivery is to be performed in conjunction with the clinically appropriate approach to collect standard of care biopsy samples to confirm disease progression. The PI has the discretion to approach via endoluminal or percutaneous method if the target(s) is/are amenable. PEF treatment will be delivered to accessible new areas of growth on existing tumors or new tumors.

Treatment may be delivered via either an endoluminal (bronchoscopic) or percutaneous approach at the discretion of the clinical investigator utilizing two available device configurations:

* Endoluminal: Galvanize Aliya System with compatible commercially available TBNA Needle and RF probe electrode
* Percutaneous: Galvanize Aliya System with compatible commercially available RF needle and RF probe electrode

The study will enroll and treat up to 30 adult patients at up to 5 clinical sites.

ELIGIBILITY:
Inclusion Criteria:

* Patient is eligible for inclusion if diagnosed and currently under physician care for one of the following advanced stage or metastatic conditions:

  * Stage IV non-small cell lung cancer
  * Stage IV hepatocellular carcinoma
  * Stage IV renal cell carcinoma
* Patient is currently receiving PD-1/PD-L1 axis immunotherapy as their most recent line of therapy, either alone or in combination with standard of care systemic therapy for their malignancy.
* Patient has exhibited at least 6 months of response to PD-1/PD-L1 axis immunotherapy regimen (defined as complete response (CR), partial response (PR), or stable disease (SD) in their index tumors per RECIST 1.1) prior to progression.
* Patient has radiologically documented or confirmed progressive disease (per RECIST 1.1) defined as a total of ≤ 5 new areas of growth on existing tumors and/or new tumors.
* New tumors must be ≤ 2cm in longest diameter. New areas of growth on existing tumors must be ≤ 2cm in longest diameter. Tumors and new areas of growth must be deemed suitable by the investigator for complete treatment with PEF. Pathologic lymph nodes must be ≥ 15mm in short axis.
* In the judgement of the investigator, the patient is able to remain on PD-1/PD-L1 axis immunotherapy for at least 3 months after PEF treatment.
* New tumors and areas of growth on existing tumors are amenable to core or forceps biopsy in order to confirm disease progression.
* Patient must be willing to undergo tumor biopsy at PEF treatment delivery.
* Patient refuses surgery and/or stereotactic body radiotherapy (SBRT).
* Life expectancy ≥ 12 weeks.
* ECOG performance status 0-1

Exclusion Criteria:

* Patient has implanted lung devices or electronic devices.
* Patient is receiving bevacizumab concurrently with their PD-1/PD-L1 axis immunotherapy.
* Patient has received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) in another study within 21 days prior to study enrollment.
* Patient is scheduled to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for off-label cancer treatment while on this study.
* Patient has unresolved adverse reaction to immunotherapy that requires dose modification.
* Patient has received any radiation therapy within 6 weeks prior to study enrollment.
* Patient has leptomeningeal disease or active brain metastases that are not clinically controlled and asymptomatic for at least 14 days following treatment and prior to study enrollment or has residual neurological dysfunction and has not been off corticosteroids for at least seven days prior to study enrollment.
* Patient has an active autoimmune disease that has required systemic treatment in past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Patient has received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within seven days prior to study enrollment. Inhaled or topical steroids, and adrenal replacement doses ≤ 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
* Patient has any history of primary immunodeficiency.
* Patient has any history of organ transplant that requires use of immunosuppressives.
* Patient has clinical signs or symptoms of active tuberculosis infection.
* Patient has history of (non-infectious) pneumonitis that required steroids or current pneumonitis/interstitial lung disease.
* Patient has documented evidence of acute hepatitis or has an active or uncontrolled infection.
* Patient has undergone major surgery within 28 days prior to study enrollment or has planned for other major surgery to be performed while enrolled in the clinical trial.
* Patient is unable or unwilling to complete all required screening and/or follow-up assessments.
* Patient is currently enrolled in another interventional clinical trial or is receiving treatment with an investigational medication or medical device that conflicts with the study protocol.
* Patient for whom the investigator considers that the PEF treatment is not in the patient's best interest.
* Patient has active alcohol or drug addiction or any other condition that, in the investigator's opinion, would interfere with their ability to comply with the study requirements.
* Patient has any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Device and Procedure serious adverse event rate | 30 days
  The rate of system-related and procedure-related serious adverse events (SAEs)
Radiologic local control | 90 days
  Frequency of radiological assessment of response of PEF-treated tumors and lymph nodes (e.g., change in longest diameter of tumor, change in short axis of lymph node)

SECONDARY OUTCOMES:
Immunologic response: lymphocytes | all time points up to 1 year
  Changes from baseline in lymphocytes (CD3+, CD4+, CD8+, Treg, NK, Neutrophils MDSC; all analyzed as cells per mL)
Immunologic response: cytokines | all time points up to 1 year
  Changes from baseline in serum levels of cytokines (IL-2, IL-6, IL-10, IL-12; all analyzed as concentration in pg / mL) from blood samples

OTHER OUTCOMES:
Procedural Success | Time of procedure
  Procedural success of accessing tumors and delivering PEF treatment
Duration of checkpoint inhibitor treatment | 12 months
  Duration of checkpoint inhibitor treatment beyond PEF treatment
Patient progression free survival (PFS) | 90 days
  Patient progression free survival (PFS)
  * PEF-treated tumor progression, new tumor appearance after PEF treatment, transition from indeterminate to cancer of previously existing lesion
Overall survival | 12 months
  Patient overall survival (OS)
Time to focal re-intervention | 12 months
  Time to focal re-intervention of PEF-treated tumor(s)

CONTACTS AND LOCATIONS:
Locations (3):
- Prince of Wales Hospital, Shatin, Hong Kong
- Radboud University Medical Center, Nijmegen, Netherlands
- Hospital Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jimenez M, Fernandez JM, Krimsky WS. Pulsed Electric Field (PEF) treatment of progressive non-small cell lung cancer concurrently treated with immune checkpoint blockade: A case report. Respir Med Case Rep. 2024 Mar 29;49:102018. doi: 10.1016/j.rmcr.2024.102018. eCollection 2024. PMID 38601720